CLINICAL TRIAL: NCT02732379
Title: Evaluating the Efficacy of Aromatherapy on Postoperative Nausea, Vomiting
Brief Title: Effect of Aromatherapy on Postoperative Nausea, Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PONV
Record Dates: First submitted 2016-03-30; First posted 2016-04-08 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; Aromatherapy; Quality of Health Care
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aromatherapy; lavender oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lavender Aromatherapy (Experimental): Aromatherapy with lavender essential oil.
  Interventions: Procedure: Lavender Aromatherapy
- Rose Aromatherapy (Experimental): Aromatherapy with rose essential oil
  Interventions: Procedure: Rose Aromatherapy
- Ginger Aromatherapy (Experimental): Aromatherapy with ginger essential oil
  Interventions: Procedure: Ginger Aromatherapy
- Placebo Aromatherapy (Placebo Comparator): Aromatherapy with pure water
  Interventions: Procedure: Placebo Aromatherapy

INTERVENTIONS:
Procedure: Lavender Aromatherapy — the two drops of lavender essential oil will be dropped into the gauze and the patient will inhale it for 5 minutes.
  Other Names: Aromatherapy with lavender essential oil
  Arms: Lavender Aromatherapy
Procedure: Rose Aromatherapy — the two drops of rose essential oil will be dropped into the gauze and the patient will inhale it for 5 minutes.
  Other Names: Aromatherapy with rose essential oil
  Arms: Rose Aromatherapy
Procedure: Ginger Aromatherapy — the two drops of ginger essential oil will be dropped into the gauze and the patient will inhale it for 5 minutes.
  Other Names: Aromatherapy with ginger essential oil
  Arms: Ginger Aromatherapy
Procedure: Placebo Aromatherapy — the two drops of pure water will be dropped into the gauze and the patient will inhale it for 5 minutes
  Other Names: Aromatherapy with pure water
  Arms: Placebo Aromatherapy

SUMMARY:
The aim of this study is to evaluate the effect of the aromatherapy with lavender, rose or ginger essential oils on nausea, vomiting and postoperative quality of recovery scores in patients with postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Postoperative Nausea and Vomiting (PONV) relief is still challenge for the anesthesiologist. Pharmacological therapies is also cornerstone for treatment of PONV. Although future researches are needed, there is some proofs about the aromatherapy could provide an inexpensive, noninvasive and effective treatment for PONV.

ELIGIBILITY:
Inclusion Criteria :

* Be scheduled for elective surgery
* Have a postoperative nausea and vomiting

Exclusion Criteria:

* Age > 65years or <18 years
* Not accepted to inhale lavender, rose or ginger oil
* Preoperative predications with anti emetic drugs
* Pregnancy or breastfeeding
* Asthma, Chronic obstructive pulmonary disease
* Poor sense of smell
* Allergy to the lavender, rose or ginger oil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-04; Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
The change of the nausea scores | During postoperative 24 hours
  Nausea will be measured with verbal descriptive scale on 0 to 3 Likert-type scale(0=no nausea, 1=some, 2= a lot, 3= severe)
The change of the vomiting score | During postoperative 24 hours
  Vomiting will be measured with verbal descriptive scale (0=no vomiting, 1= 1 time, 2= 2 or 3 times, 3= 4 times and up)

SECONDARY OUTCOMES:
The consumption of the antiemetic drug | During postoperative 24 hours
  The antiemetic drug dose will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Karaman, MD, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University Medical School Hospital, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided